CLINICAL TRIAL: NCT00669786
Title: Highly Purified Human Menopausal Gonadotropin Versus Recombinant Follicle Stimulating Hormone in Ovarian Hyperstimulation With Gonadotropin Releasing Hormone Antagonists. A Randomized Study.
Brief Title: Human Menopausal Gonadotropin (HMG) vs Recombinant Follicle Stimulating Hormone (rFSH) in Gonadotropin Releasing Hormone (GnRH) Antagonist Cycles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Other Study IDs: VLC-EB-0103-0408-1
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2008-05-01 (Estimated); Status verified 2008-04

CONDITIONS: Ovarian Stimulation
Keywords: Ongoing Pregnancy Rate
MeSH Terms: interventions — Menotropins; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HMG (Active Comparator): Human Menopausal Gonadotropin (HMG)
  Interventions: Drug: Human Menopausal Gonadotropin (HMG) & - Recombinant Follicle Stimulating Hormone (r-FSH)
- r-FSH (Active Comparator): Recombinant Follicle Stimulating Hormone
  Interventions: Drug: Human Menopausal Gonadotropin (HMG) & - Recombinant Follicle Stimulating Hormone (r-FSH)

INTERVENTIONS:
Drug: Human Menopausal Gonadotropin (HMG) & - Recombinant Follicle Stimulating Hormone (r-FSH)

SUMMARY:
A randomized controlled trial comparing the ongoing pregnancy rate (primary end-point) in 280 patients undergoing IVF/ICSI after stimulation with hp-hMG or rFSH controlled with a GnRH antagonist. Non significant differences were observed between hp-hMG and rFSH in terms of the ongoing pregnancy rate per started cycle (35.0% vs. 32.1%; p=0.61); R.R: 1.09 (95% CI: 0.78-1.51; Risk Difference: 2.9%). No differences were observed for implantation, clinical pregnancy and pregnancy loss rates. Patients receiving rFSH obtained more oocytes (14.4 ± 8.1 vs. 11.3 ± 6.0; p=0.001). Estradiol was higher at the end of stimulation in the hp-hMG group, while Progesterone was higher in patients stimulated with rFSH.

ELIGIBILITY:
Inclusion Criteria:

* women with good physical and mental health
* aged 18-37 years
* regular menstrual cycles ranging from 25 to 35 days; body mass index (BMI) < 30 kg/m2
* normal basal serum FSH (≤ 10 IU/L) and E2 (≤ 75 pg/mL) levels determined on the day 3 of the cycle previous to COH
* no uterine (fibroids, adenomyosis, mullerian malformations), ovarian (endometrioma, polycystic ovaries) or adnexa (hydrosalpinx) abnormalities assessed by vaginal ultrasound.

Exclusion Criteria:

* patients with a history of recurrent pregnancy loss
* any significant systemic disease, endocrine or metabolic disorder
* having concomitant medication interfering with the purposes of the study
* patients who have received any ovulation induction drug within one month before their inclusion in the study.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Spain

REFERENCES:
- [Derived] Bosch E, Vidal C, Labarta E, Simon C, Remohi J, Pellicer A. Highly purified hMG versus recombinant FSH in ovarian hyperstimulation with GnRH antagonists--a randomized study. Hum Reprod. 2008 Oct;23(10):2346-51. doi: 10.1093/humrep/den220. Epub 2008 Jun 25. PMID 18583332